CLINICAL TRIAL: NCT05065853
Title: Urinary and Vaginal HPV Testing as a Novel Cervical Cancer Screening Tool: a Diagnostic Test Accuracy Study
Brief Title: Urinary and Vaginal HPV Testing in Cervical Cancer Screening
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Aarhus (Other)
Collaborators: University Clinic for Cancer Screening, Department of Public Health Programmes, Randers Regional Hospital, Denmark (Unknown); Centre for the Evaluation of Vaccination, Vaccine & Infectious Disease Institute, Faculty of Medicine and Health Sciences, University of Antwerp, Belgium (Unknown); Department of Gynecology, Randers Regional Hospital, Denmark (Unknown); Departement of Pathology, Randers Regional Hospital , Denmark (Unknown)
Responsible Party: Principal Investigator, Mette Tranberg Nielsen, post doc, PhD, MScH, biomedical laboratory scientist, University of Aarhus
Other Study IDs: 2703
Record Dates: First submitted 2021-10-01; First posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Uterine Cervical Neoplasms
Keywords: HPV DNA tests, self-collection, cervical cancer screening
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — First-void urine samples Vaginal self-samples Clinician-collected cervical samples Cervical biopsy Cone biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: urine self-sampling group — collection of urine and vaginal samples
  Other Names: vaginal self-sampling group
Diagnostic Test: clinician-collected cervical sample group — A clinician takes a smear from cervix according to standard routine

SUMMARY:
Cervical cancer, caused by high-risk human papillomavirus (HPV) infection, poses a problem worldwide as it is the fourth most common female cancer. Fifty percent of all invasive cervical cancers occur among the 25% not attending cervical cancer screening. To reach these women, this project will contribute to the development of a novel and accurate urinary and vaginal screening tool, which allows women to collect the screening samples at home. This project tests the hypotheses: 1) urinary HPV testing is non-inferior to HPV testing on clinician-collected cervical samples for detection of high-grade cervical pre-cancer, 2) Vaginal HPV testing is non-inferior to HPV testing on clinician-collected cervical samples for detection of high-grade cervical pre-cancer and 3) DNA methylation testing is suitable as a colposcopy triage test among women with HPV-positive urine and/or vaginal samples to prevent unnecessary colposcopies and overtreatment of women without clinically meaningful HPV infections. If confirmed, urinary and vaginal HPV testing could revolutionize todays screening programs and keep Denmark at the forefront of cervical cancer prevention.

DETAILED DESCRIPTION:
Paired urine, vaginal, and clinician-collected cervical samples will be obtained from approximately 330 women aged 23-64 years referred for colposcopy and cervical biopsies due to abnormal screening result or referred for cervical excision due to treatment of CIN2+. Upon informed consent, the women will collect a first-void urine sample and a vaginal self-sample. Before colposcopy or excision, a clinician will collect a cervical sample. Among women referred for colposcopy, four cervical punch biopsies will be taken. For women referred for excision, a cone biopsy will be taken using a loop electrosurgical excision procedure. Upon arrival in the laboratory, the paired urine, vaginal and cervical samples will be HPV tested using the Cobas 4800 HPV DNA assay. Histological results will served as reference and be grouped as ≤CIN1 (normal tissue, CIN1) versus CIN2+. The performance of the six individual methylation markers and combinations thereof will be evaluated using the histological results as reference.

The primary endpoint will be the relative sensitivity and specificity of HPV testing in first-void urine, vaginal self-sample versus clinician-collected cervical samples to detect CIN2+. Non-inferiority of HPV testing between sample types will be evaluated against a margin of 90% for sensitivity and 98% for specificity. The performance of each methylation marker will be illustrated by ROC curves and assessed by the area under the curve.

ELIGIBILITY:
Inclusion Criteria:

* Females
* Aged 23-64 years
* Referred for colposcopy and cervical biopsies or referred for cervical excision

Exclusion Criteria:

* younger than 23 years
* older than 64 years
* not provided informed conte

Ages: 23 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only female can be diagnosed with cervical cancer or its precancer lesion, thus only women are candidates for inclusion.
Study Population: women aged 23-64 years referred for colposcopy and cervical biopsies due to abnormal cervical cancer screening result or referred for cervical excision due to treatment of CIN2+
Sampling Method: Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2021-10-18 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
relative sensitivity and specificity of urinary sampling | at baseline
  The primary endpoint will be the relative sensitivity and specificity of HPV testing in first-void urine versus clinician-collected cervical samples to detect CIN2+
relative sensitivity and specificity of vaginal self-sampling | at baseline
  The primary endpoint will be the relative sensitivity and specificity of HPV testing in vaginal self-samples versus clinician-collected cervical samples to detect CIN2+

CONTACTS AND LOCATIONS:
Overall Officials: Mette Tranberg, post doc, Principal Investigator — Randers Regional Hospital and Aarhus University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tranberg M, Van Keer S, Jensen JS, Norgaard P, Gustafson LW, Hammer A, Bor P, Binderup KO, Blach C, Vorsters A. High-risk human papillomavirus testing in first-void urine as a novel and non-invasive cervical cancer screening modality-a Danish diagnostic test accuracy study. BMC Med. 2025 Jun 2;23(1):327. doi: 10.1186/s12916-025-04149-0. PMID 40457337